CLINICAL TRIAL: NCT03978338
Title: A Multi-center, Randomized, Double-blind, Controlled Study to Evaluate the Efficacy and Safety of Brain Polypeptide Solution in Improving Cognitive Function in Mild Alzheimer's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Brain Polypeptide Solution in Mild Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Zhitong Biopharma CO.,LTD (Unknown)
Responsible Party: Principal Investigator, Wei Chen, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-1959
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Brain polypeptide
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group will take the brain polypeptide solution .
  Interventions: Dietary Supplement: brain polypeptide solution
- Control group (Placebo Comparator): The control group was treated with the same package of placebo .
  Interventions: Other: same package of placebo

INTERVENTIONS:
Dietary Supplement: brain polypeptide solution — The experimental group will take the brain polypeptide solution 60ml per day which contains nitrogen 90mg, soybean oil ,glycerin and soybean phospholipids in 84days.
  Arms: Intervention group
Other: same package of placebo — The control group was treated with the same package of placebo 60ml per day which contains soybean oil ,glycerin and soybean phospholipids in 84 days.
  Arms: Control group

SUMMARY:
In recent years, reduced levels of brain-derived neurotrophic factor (BDNF) have been found in dementia patients. BDNF reduces amyloid precursor protein (APP) fragments via the Trk signaling pathway, and the expression of transgenic BDNF in animal models of Alzheimer's Disease（AD）shows a protective effect on neurodegeneration. A lot of researches have proved that brain hydrolysate injection can improve the level of BDNF in the brain. And oral brain peptide dietary supplements, which is also derived from brain proteolytic products, may also adjust and improve neuron metabolism, promote the formation of synapses, induce the differentiation of neurons, and protect nerve cells from ischemia and neurotoxin damage, reduce the risk of loss of cognitive function in the aging process. However, there are still no studies on dietary supplements derived from brain protein hydrolysates in China. Therefore, the investigators designed a randomized controlled double-blind study program to preliminarily evaluate the efficacy, safety and possible mechanism of brain polypeptide solution in improving the cognition of mild alzheimer's disease patients.

The research is a prospective, multicenter, cohort study. 200 patients with mild alzheimer's disease will be selected and randomly divided into experimental group and control group according to the numerical random table. The experimental group will take the brain polypeptide solution 60ml per day and the control group was treated with the same package of placebo 60ml per day. The treatment regimen remained unchanged during the observation period. During the study period, safety index including blood and urine routine, liver and kidney function, coagulation index and clinical effect index about neuropsychological scales will be recorded.

DETAILED DESCRIPTION:
The investigators design a prospective, multicenter, cohort study.200 patients with mild Alzheimer's disease will be selected and divided into brain polypeptide nutrient solution group (experimental group) and control group according to the numerical random table. The experimental group will take brain polypeptide solution 60ml per day, while the control group took placebo in the same package 60ml per day. The observation period is 84 days. And follow-up will take place at 42 and 84 days .The treatment regimen remained unchanged during the observation period. Safety indexes include blood and urine routine, liver and kidney function, coagulation index, etc. Screening indexes include syphilis antibody, HIV antibody, hepatitis b virus antibody, hepatitis c virus antibody, folic acid, vitamin B12, etc. Clinical outcome indicators include a number of scales to evaluate neurological and cognitive functions, such as the Alzheimer's disease assessment scale-cognitive subscale (ADAS-cog). Mechanism related indicators such as metabolomics was used to understand the possible differences in metabolic indicators. It is helpful to guide the use of brain polypeptide in Alzheimer's patients correctly .

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 50 to 85 (including 50 and 85 years old), regardless of ethnic group or gender;
2. The subjects should be able to complete the cognitive ability measurement and other tests specified in the protocol;
3. meeting the criteria for likely Alzheimer's Disease （AD） dementia (2007) by National Institute of Neurological Disorders and Strokes - Alzheimer's Disease and Related Diseases Association（NINCDS-ADRDA）;
4. patients with mild dementia: the total score of Mini-Mental State Examination (MMSE) : illiteracy ≤17 points, primary school ≤20 points, secondary school ≤22 points, university ≤23 points; Clinical Dementia Rating scale （CDR） = 1 point;
5. the total score of the Hachinski Ischemic Score （HIS ）was < 4.
6. Hamilton depression scale (17 items) total score ≤7 points;
7. Brain MRI shows a high likelihood of AD;
8. before enrollment, patients should take a stable dose of dementia drugs (such as donepezil 10mg) ≥8 weeks;
9. the expected survival time is > 1 year;
10. subjects should have a stable and reliable caregiver, or at least have frequent contact with the caregiver (at least 3 days per week and at least 2 hours per day), who will help patients participate in the whole study; Caregivers must accompany the subjects to the visit and assist in completing the relevant scale.

Exclusion Criteria:

1. refuse to sign the inform consent form;
2. other causes of dementia: known vascular, central nervous system infection ,Parkinson's disease, traumatic brain dementia, other physical and chemical factors; serious body disease , intracranial space-occupying lesions, endocrine system disease, such as thyroid disease, and a lack of vitamin B12, folic acid, or any other known causes of dementia.
3. central nervous system diseases (including stroke, optic neuromyelitis, Parkinson's disease, epilepsy, etc.);
4. obvious positive signs of nervous system examination;
5. psychotic patients, including schizophrenia or other disorders with bipolar disorder, major depression or delirium;
6. uncontrolled hypertension or hypotension during screening: systolic blood pressure ≥180（millimetres of mercury ）mmHg or < 90mmhg, or diastolic blood pressure ≥120mmHg or < 60mmhg;
7. unstable or severe diseases of the heart, lung, liver, kidney and hematopoietic system according to the judgment of the researchers;
8. patients with incurable visual and auditory disorders that cannot complete neuropsychological tests and scales;
9. female subjects who are positive in pregnancy test or breast-feeding and who cannot take effective contraceptive measures or have a birth plan;
10. severe allergy, non-allergic drug reaction or multi-drug allergy history;
11. participated in other clinical trials within 3 months before screening visit;
12. taking any health care products related to brain and brain improvement currently and failing to keep the promise to stop using the above products;
13. other conditions are unsuitable for participating in this study according to the judgement of researchers.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Changes of Alzheimer's Disease Assessment Scale-Cognitive Subscale(ADAS-cog) scores | baseline time,week 12.
  ADAS-cog will be performed to test the cognition of patients at the enrollment and week 12.The score ranges from 0 to 75，and higher values represent a better outcome.

SECONDARY OUTCOMES:
Changes of Alzheimer's Disease Collaborative research group-Activities of Daily Living(ADCS-ADL)scores | baseline time,week6,week 12.
  ADCS-ADL will be performed to test the activities of patients at the enrollment,week 6 and week12.The score ranges from 0 to 54，and higher values represent a better outcome.
Changes of Pittsburgh sleep quality index (PSQI) scores | baseline time,week6,week 12.
  PSQI will be performed to test the sleep quality of patients at the enrollment ,week 6 and week12.The score ranges from 0 to 21，and higher values represent a worse outcome.
Changes of Neuropsychiatric Inventory(NPI )scores | baseline time,week 12.
  NPI will be performed to test the mental symptoms of patients at the enrollment and week12.The score ranges from 0 to 144，and higher values represent a worse outcome.
Changes of ( Mini-Mental State Examination )MMSE scores | baseline time,week 12.
  MMSE will be performed to test the cognition of patients at the enrollment and week12.The score ranges from 0 to 30，and higher values represent a better outcome.
Changes of Montreal Cognitive Assessment (MoCA) scores | baseline time,week 12.
  MoCA will be performed to test the cognition of patients at the enrollment and week12.The score ranges from 0 to 30，and higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, M.D., Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Yes
The following data will be shared at the end of the study: demographic data, current medical history, past history,physical examination data and date of neuropsychological evaluation collected at this research.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data is expected to be available after,September, 2020 and can be used forever.
Access Criteria: The information should be used for academic research, medical communication, etc., and is prohibited from being used for commercial gain.

REFERENCES:
- [Background] McEvoy CT, Guyer H, Langa KM, Yaffe K. Neuroprotective Diets Are Associated with Better Cognitive Function: The Health and Retirement Study. J Am Geriatr Soc. 2017 Aug;65(8):1857-1862. doi: 10.1111/jgs.14922. Epub 2017 Apr 25. PMID 28440854
- [Background] Kmietowicz Z. Mediterranean diet is associated with reduced brain shrinkage in older people, study finds. BMJ. 2015 Oct 21;351:h5556. doi: 10.1136/bmj.h5556. No abstract available. PMID 26493230
- [Background] Alvarez XA, Cacabelos R, Laredo M, Couceiro V, Sampedro C, Varela M, Corzo L, Fernandez-Novoa L, Vargas M, Aleixandre M, Linares C, Granizo E, Muresanu D, Moessler H. A 24-week, double-blind, placebo-controlled study of three dosages of Cerebrolysin in patients with mild to moderate Alzheimer's disease. Eur J Neurol. 2006 Jan;13(1):43-54. doi: 10.1111/j.1468-1331.2006.01222.x. PMID 16420392
- [Background] Gauthier S, Proano JV, Jia J, Froelich L, Vester JC, Doppler E. Cerebrolysin in mild-to-moderate Alzheimer's disease: a meta-analysis of randomized controlled clinical trials. Dement Geriatr Cogn Disord. 2015;39(5-6):332-47. doi: 10.1159/000377672. Epub 2015 Mar 26. PMID 25832905
- [Background] Alvarez XA, Cacabelos R, Sampedro C, Couceiro V, Aleixandre M, Vargas M, Linares C, Granizo E, Garcia-Fantini M, Baurecht W, Doppler E, Moessler H. Combination treatment in Alzheimer's disease: results of a randomized, controlled trial with cerebrolysin and donepezil. Curr Alzheimer Res. 2011 Aug;8(5):583-91. doi: 10.2174/156720511796391863. PMID 21679156
- [Background] Muresanu DF, Alvarez XA, Moessler H, Buia M, Stan A, Pintea D, Moldovan F, Popescu BO. A pilot study to evaluate the effects of Cerebrolysin on cognition and qEEG in vascular dementia: cognitive improvement correlates with qEEG acceleration. J Neurol Sci. 2008 Apr 15;267(1-2):112-9. doi: 10.1016/j.jns.2007.10.016. Epub 2007 Nov 28. PMID 18048059